CLINICAL TRIAL: NCT06992856
Title: The Effect of Cap-assisted Water Exchange Colonoscopy on Straight Passage of the Colonoscope Through the Sigmoid Colon, Without Loop Formation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhijun Bao, Director, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2025K235
Record Dates: First submitted 2025-05-20; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Colonoscope Passage
Keywords: colonoscope passage; left colon water exchange; cap-assisted; without loop formation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- conventional colonoscope passage (Active Comparator): Use conventional colonoscope passage through the sigmoid colon
  Interventions: Procedure: Conventional colonoscope passage
- left colon water exchange colonoscope passage (Experimental): Use left colon water exchange colonoscope passage through the sigmoid colon
  Interventions: Procedure: left colon water exchange colonoscope passage
- Cap-assisted left colon water exchange colonoscope passage (Experimental): Use Cap-assisted left colon water exchange colonoscope passage through the sigmoid colon
  Interventions: Procedure: cap-assisted left colon water exchange colonoscope passage

INTERVENTIONS:
Procedure: Conventional colonoscope passage — Use conventional colonoscope passage through the sigmoid colon
  Arms: conventional colonoscope passage
Procedure: left colon water exchange colonoscope passage — Use left colon water exchange colonoscope passage through the sigmoid colon
  Arms: left colon water exchange colonoscope passage
Procedure: cap-assisted left colon water exchange colonoscope passage — Use cap-assisted left colon water exchange colonoscope passage through sigmoid colon
  Arms: Cap-assisted left colon water exchange colonoscope passage

SUMMARY:
A prospective, single-center, single-blind, randomized controlled study to compare the proportion of straight passage through the sigmoid colon without loop formation between conventional colonoscope passage, left colon water exchange colonoscope passage, and cap-assisted left colon water exchange colonoscope passage through the sigmoid colon

DETAILED DESCRIPTION:
1. Patients are undergone screening, surveillance, or therapeutic colonoscopy at the Endoscopy department of Gastrointestinal endoscopy center of Huadong hospital affiliated to Fudan University.
2. Randomize patients into 3 interventional groups based on R script (version 4.4.1), including (1) Group 1: Conventional colonoscope passage, (2) Group 2: left colon water exchange colonoscope passage, (3) Group 3: cap-assisted left colon water exchange colonoscope passage.
3. Collecting variables which consist of primary and secodary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-80 years
* sedation colonoscopy

Exclusion Criteria:

* History of colorectal surgery
* Clinical suspicion of, or pathologically confirmed, colorectal cancer
* Presence of any "alarm" symptom or sign-hematochezia, melena, unexplained anemia or weight loss, palpable abdominal mass, or a positive digital rectal examination
* Pregnancy or lactation
* Known or suspected gastrointestinal obstruction
* Diagnosed inflammatory bowel disease
* Use of antiplatelet or anticoagulant therapy (e.g., aspirin, warfarin) within 7 days before colonoscopy or any documented coagulation disorder
* Current enrolment in another clinical study or participation in any clinical trial within the previous 60 days
* Requirement for emergency colonoscopy
* Any other condition that, in the investigators' judgment, renders the patient unsuitable for inclusion in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 531 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of straight passage through the sigmoid colon without loop formation | immediately after the procedure

SECONDARY OUTCOMES:
Cecal intubation rate | immediately after the procedure
Cecal intubation time | immediately after the procedure
Time of insertion to cecum | immediately after the procedure
Colonoscope insertion failure rate | immediately after the procedure
Adenoma detection rate | 2 weeks after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Danian Ji, M.D., Study Director — Huadong Hospital
Locations (1):
- Huadong hospital affiliated to Fudan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1 year after completion of this study
Access Criteria: All researchers can require the original data from principal investigator of this study (Email address: arctg4@163.com)